CLINICAL TRIAL: NCT03415867
Title: A Phase 1b/ 2a Pilot Trial of the Oral Hedgehog Signalling Inhibitor Glasdegib in Patients With Sclerotic Chronic Graft-Versus-Host Disease Refractory to Second-Line Treatment
Brief Title: Glasdegib in Refractory Patients With Sclerotic Chronic Graft-Versus-Host Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Grupo Espanol de trasplantes hematopoyeticos y terapia celular (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GLAS; 2017-000862-31 (EudraCT Number)
Record Dates: First submitted 2017-12-05; First posted 2018-01-30 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Sclerodermoid Chronic Graft-Versus-Host Disease (Disorder)
Keywords: Graft-versus-host disease; Bone marrow transplantation; Hedgehog inhibitor
MeSH Terms: conditions — Graft vs Host Disease | interventions — glasdegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation sequential cohorts (Experimental): Glasdegib will be self-administered orally once daily in the morning as monotherapy in continuous 28-day treatment cycles for a maximum of 24 cycles. Those patients enrolled in the trial that obtain objective clinical benefit under treatment with glasdegib (defined as the achievement of at least a partial response at one or more target organs), will be allowed to proceed to a slow dose withdrawal phase over a period of 6 months after the end of Cycle 24. The dose reduction scheme is fully detailed in the protocol.
  Interventions: Drug: Glasdegib

INTERVENTIONS:
Drug: Glasdegib — A dose escalation/de-escalation design will be applied in successive patient cohorts until identification of MTD (dose range: 25-200 mg OD).
  Other Names: PF-04449913

SUMMARY:
This is a phase 1b/2a, open label, multi-centre, safety and efficacy study of glasdegib in patients with sclerotic cGVHD refractory to second-line treatment. The design for the current study is a standard 3+3 dose-finding scheme. A dose escalation/de-escalation design will be applied in successive patient cohorts until identification of MTD. Glasdegib will be self-administered orally once daily in the morning as monotherapy in continuous 28-day treatment cycles for a maximum of 24 cycles. Those patients enrolled in the trial that obtain objective clinical benefit under treatment with glasdegib (defined as the achievement of at least a partial response at one or more target organs), will be allowed to proceed to a slow dose withdrawal phase over a period of 6 months after the end of Cycle 24.

DETAILED DESCRIPTION:
Three patients will be initially treated at the corresponding dose level of glasdegib at each dose escalation stage. Dose escalation will be started in a first cohort of 3 patients at a starting dose of 50 mg (Dose Level 1) and will then proceed as follows:

* If no dose-limiting toxicity is observed among the first 3 patients in a cohort, then 3 additional patients will be treated at the next higher dose level.
* If a dose-limiting toxicity is observed in 1 of the initial 3 treated patients, 3 additional patients, resulting in a total of 6 patients, will be enrolled and treated at the same dose level.
* If no further dose-limiting toxicity is observed (1/6 patients), dose escalation will continue to the next dose level in a new cohort of 3 patients.
* If ≥ 2/3 or 2/6 patients experience a dose-limiting toxicity, then MTD has been exceeded and the next lower dose of glasdegib will be expanded until a total number of 6 patients treated at that dose level is reached. If 0 or 1 patient out of 6 experiences a dose-limiting toxicity, this dose level will be declared MTD. If ≥ 2/6 patients experience a dose-limiting toxicity, the next lower dose level will be expanded.
* Prior safety data evaluation and approval by an independent data monitoring committee will be required before escalation at each dose level.

In case that MTD is exceeded within the first cohort, then a -1 Dose Level (25 mg OD) will be tested. If MTD is exceeded at 25 mg OD, the trial will be stopped and no additional testing of glasdegib at lower doses will be allowed.

Dose escalation will continue following the above-specified rules until MTD is declared. Once MTD is defined, dose expansion at MTD in cohorts of 3 patients will proceed until the pre-established sample size (20 patients) is reached. In the event that the highest pre-defined dose (200 mg OD) is tested in two successive cohorts of 3 patients and MTD is not attained, dose expansion at 200 mg OD will precede until a sample size of 20 patients is reached. The administered dose level may be subject to further adjustment (dose reduction only) in the dose expansion phase based on emerging safety, pharmacokinetic or pharmacodynamic data.

Additional dose levels may be explored, if appropriate, based on emerging safety, pharmacokinetic, or pharmacodynamic data, prior safety data evaluation and approval by an external monitoring committee.

Patients who are not evaluable for dose-limiting toxicity (e.g., those not receiving at least 80% of the planned dose of glasdegib in the dose-limiting toxicity monitoring period (first 2 cycles) for reasons other than study treatment-related toxicities) must be replaced.

If the pre-specified sample size is completed before MTD is defined or before the highest pre-defined dose (200 mg OD) is tested in at least 6 patients, additional patients may be recruited into the study (for a total sample size of up to 24 patients) until MTD is defined or two cohorts of 3 patients complete treatment at 200 mg OD.

Glasdegib may be dose reduced or discontinued during any cycle based on the patient's individual tolerability. During the dose-escalation phase, once a patient has a dose reduction for a study drug-related toxicity; the dose will not be re-escalated. Dose re-escalation up to the MTD will be allowed at the investigator's discretion during the dose expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥ 18 years old) recipients of an allogeneic hematopoietic stem cell transplantation with active sclerotic cGVHD without response, in partial response or in relapse after 2 previous lines of treatment including corticosteroids and one of the following second line treatments:

   * Extracorporeal photopheresis (preferably).
   * A calcineurin inhibitor.
   * A mammalian target of rapamycin (mTOR) inhibitor.
   * Pentostatin.
   * Rituximab.
   * Imatinib.
   * Ruxolitinib.
2. Eastern Cooperative Oncology Group Performance Status 0 to 2.
3. Adequate organ function as defined by the following:

   * Serum aspartate aminotransferase (AST) and serum alanine aminotransferase (ALT) ≤ 3 x upper limit of normal (ULN).
   * Total serum bilirubin ≤ 2 x ULN (except patients with documented Gilbert's syndrome).
   * Serum creatinine ≤ 1.5 x ULN or estimated creatinine clearance ≥ 60 mL/min as calculated using the method standard for the institution.
4. Hematologic malignancy in complete remission.
5. Resolved acute effects of any prior therapy to baseline severity or Grade ≤ 1 CTCAE except for adverse events not constituting a safety risk by investigator judgement.
6. Serum/urine pregnancy test (for females of childbearing potential) that is negative at screening and immediately prior to initiation of treatment (first dose). Male and female patients of childbearing potential must agree to use highly effective methods of contraception throughout the study and for at least 180 days after the last dose of assigned treatment. A patient is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active.
7. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legal representative) has been informed of all pertinent aspects of the study.
8. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures.

Exclusion Criteria:

Patients presenting with any of the following will not be included in the study:

1. Patients with active malignancy with the exception of basal cell carcinoma, nonmelanoma skin cancer or cervical carcinoma-in-situ. Other prior or concurrent malignancies will be considered on a case-by-case basis.
2. Any one of the following, currently or in the previous 6 months: myocardial infarction, congenital long QT syndrome, torsade de pointes or clinically significant ventricular arrhythmias.
3. QTc interval >470 milliseconds using the Fridericia (QTcF).
4. Patients with an active, life threatening or clinically significant uncontrolled systemic infection.
5. Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness or active Hepatitis B or C infection.
6. Known malabsorption syndrome or other condition that may impair absorption of study medication (e.g., gastrectomy or lap band).
7. Major surgery or radiation within 4 weeks of starting study treatment.
8. Prior treatment with:

   * A hedgehog inhibitor at any time.
   * An investigational agent for the treatment of cGVHD (a three-month wash-out period will be required).
9. Concurrent treatment with any investigational agent.
10. Concurrent administration of herbal preparations.
11. Current use at time of study entry or anticipated need for drugs that are known strong CYP3A4/5 inducers.
12. Current drug or alcohol abuse.
13. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
14. Patients who are investigational site staff members or relatives of those site staff members directly involved in the conduct of the trial.
15. Pregnant females; breastfeeding females; males and females of childbearing potential not using two methods of highly effective contraception or not agreeing to continue two methods of highly effective contraception for at least 180 days after last dose of investigational product.
16. Recent or active suicidal ideation or behaviour.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2022-01-09 (Actual); Study Completion 2022-06-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose. | Up to 48 weeks.
  To determine the maximum tolerated dose (MTD) or maximum administered dose (MAD) and/or the recommended Phase 2 dose (RP2D) of glasdegib in subjects with sclerotic cGVHD.

SECONDARY OUTCOMES:
Adverse events. | Adverse events will be assessed from the date the informed consent document is signed until 28 days after the last administered dose of glasdegib.
  Type, incidence, severity (graded by the National Cancer Institute [NCI] Common.
  Terminology Criteria for Adverse Events [CTCAE], Version 4.0), timing, intensity, and relatedness of adverse events.
Overall response rate (ORR). | Response to treatment will be evaluated on Day 1 of Cycles 1, 2, 4, 7, 10, 13, 16, 19, 22, 25, 28 (each cycle is 28 days) and end treatment.
  ORR as assessed by the NIH cGVHD Response Criteria.
Immunosuppression requirements. | Modifications to the immunosuppressive regimen will be assessed from date of study entry to study withdrawal or end of treatment (up to 48 weeks).
  Dose reduction and/or withdrawal of concomitantly administered immunosuppressive drugs.
Duration of clinical response. | Response to treatment will be evaluated on Day 1 of Cycles 1, 2, 4, 7, 10, 13, 16, 19, 22, 25, 28 (each cycle is 28 days) and day 28 of Cycle 24,
  Duration of clinical response as assessed by the NIH cGVHD Response Criteria.
Survival outcomes: overall survival. | Survival status of participants will be followed from inclusion to end of trial (once every recruited patient has completed 12 cycles of treatment or withdrawn from the study).
  Overall survival (OS).
Survival outcomes: progression-free survival. | Progression-free survival status of participants will be followed from inclusion to end of trial (once every recruited patient has completed 12 cycles of treatment or withdrawn from the study).
  Progression-free survival (PFS).
Pharmacokinetics: elimination half-life. | Day 1 of Cycles 1, 2 and 4 (each cycle is 28 days).
  Elimination half-life of glasdegib.
Pharmacokinetics: AUC. | Day 1 of Cycles 1, 2 and 4 (each cycle is 28 days).
  Area under the plasma concentration versus time curve (AUC) for each dose group.
Pharmacokinetics: Cmax. | Day 1 of Cycles 1, 2 and 4 (each cycle is 28 days).
  Maximum plasma concentration (Cmax) for each dose group.
Pharmacodynamics: Gli1 expression. | Day 1 of Cycle 1 and Cycle 2, 4 , 13 and 25 (or End of Treatment if the patient does not subsequently proceed to the dose reduction phase) .
  To explore the relationship of glasdegib plasma levels and Gli1 expression in peripheral blood mononuclear cells.
Pharmacodynamics: Gli2 expression | Day 1 of Cycle 1 and Cycle 2, 4 , 13 and 25 (or End of Treatment if the patient does not subsequently proceed to the dose reduction phase) .
  To explore the relationship of glasdegib plasma levels and Gli2 expression in peripheral blood mononuclear cells.
Pharmacodynamics: Shh expression. | Day 1 of Cycle 1 and Cycle 2, 4 , 13 and 25 (or End of Treatment if the patient does not subsequently proceed to the dose reduction phase) .
  To explore the relationship of glasdegib plasma levels and Shh expression in peripheral blood mononuclear cells.

CONTACTS AND LOCATIONS:
Overall Officials: José Antonio Pérez-Simón, M.D. Ph.D., Study Chair — Department of Hematology, Hospital Universitario Virgen del Rocío. Spain
Locations (6):
- Spain (6):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data for primary and secondary variables is planned to be shared with all participants within 6 months of data completion
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after data completion
Access Criteria: Investigators participating in the study until the final publication is done

REFERENCES:
- [Background] Inamoto Y, Storer BE, Petersdorf EW, Nelson JL, Lee SJ, Carpenter PA, Sandmaier BM, Hansen JA, Martin PJ, Flowers ME. Incidence, risk factors, and outcomes of sclerosis in patients with chronic graft-versus-host disease. Blood. 2013 Jun 20;121(25):5098-103. doi: 10.1182/blood-2012-10-464198. Epub 2013 Apr 1. PMID 23547053
- [Background] Dignan FL, Amrolia P, Clark A, Cornish J, Jackson G, Mahendra P, Scarisbrick JJ, Taylor PC, Shaw BE, Potter MN; Haemato-oncology Task Force of British Committee for Standards in Haematology; British Society for Blood and Marrow Transplantation. Diagnosis and management of chronic graft-versus-host disease. Br J Haematol. 2012 Jul;158(1):46-61. doi: 10.1111/j.1365-2141.2012.09128.x. Epub 2012 Apr 26. PMID 22533811
- [Background] Zerr P, Palumbo-Zerr K, Distler A, Tomcik M, Vollath S, Munoz LE, Beyer C, Dees C, Egberts F, Tinazzi I, Del Galdo F, Distler O, Schett G, Spriewald BM, Distler JH. Inhibition of hedgehog signaling for the treatment of murine sclerodermatous chronic graft-versus-host disease. Blood. 2012 Oct 4;120(14):2909-17. doi: 10.1182/blood-2012-01-403428. Epub 2012 Aug 22. PMID 22915638